CLINICAL TRIAL: NCT04949074
Title: Collection of SARS-CoV-2 RNA Extracted From Nasopharyngeal and Saliva Samples From Same Patients
Brief Title: Collection of RNA Extracted From Nasopharyngeal and Saliva Samples From Same Patients With Suspicion of Covid-19
Acronym: COLL001
Status: Completed | Type: Observational
Sponsor: ID Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-A00877-34
Record Dates: First submitted 2021-06-22; First posted 2021-07-02 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2022-04

CONDITIONS: Respiratory Tract Infections
Keywords: SARS-CoV-2; saliva; diagnostic
MeSH Terms: conditions — Respiratory Tract Infections; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — RNA extracted from nasopharyngeal and saliva / sputum extracts from the same patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- RNA extracted from Positive NSP samples: RNA extracted from NSP samples, found positive for the presence of SARS-CoV-2
- RNA extracted from Positive saliva samples: RNA extracted from saliva samples found positive for the presence of SARS-CoV-2
  Interventions: Other: saliva sampling
- RNA extracted from negative NSP samples: RNA extracted from NSP samples, found negative for the presence of SARS-CoV-2
- RNA extracted from negative saliva samples: RNA extracted from saliva samples found negative for the presence of SARS-CoV-2
  Interventions: Other: saliva sampling

INTERVENTIONS:
Other: saliva sampling — when the patient goes to the laboratory for a covid 19 diagnostic from a routine nasopharingeal sample, an additionnal sample of saliva is asked
  Groups: RNA extracted from Positive saliva samples; RNA extracted from negative saliva samples

SUMMARY:
Constitution of a collection of SARS-CoV-2 RNA extracts from nasopharyngeal and saliva / sputum samples, from the same patients (paired samples), taken during the same consultation in an indication of detection of SARS-CoV-2 in with a view to developing tests / diagnostic tools for SARS-CoV-2.

DETAILED DESCRIPTION:
In order to preserve their anonymity, the participant will be identified in a dedicated form by a unique identification number. An identification list of participants will be kept in the investigator's file. The investigator will ensure that the anonymity of each person participating in the research is guaranteed.

The source documents are the original documents, data and files from which the data concerning the participant is reported in the Data set_COLL001.xls form provided to the investigator which will serve as an observation notebook.

The investigator must agree to allow direct access to research source data during monitoring, audit or inspection visits. The source data is for the most part computerized and accessible after authorization.

The data will be transcribed into an Excel form Data set_COLL001.xls pseudonymized form which will serve as an observation book. The data will be recorded and then transmitted to ID SOLUTIONS via the Data set_COLL001.xls form provided to the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Male, female adult
* Patient with an indication for SARS-CoV-2 screening.
* Patient having been informed and having given his non-objection to participate in the study
* Patient affiliated with a French social security scheme or beneficiary of such a scheme

Exclusion Criteria:

* Pregnant or breastfeeding women
* Vulnerable people Adults placed under tutorship or curatorship or under judicial protection, Patient unable to personally give consent, or adult protected by law, Opposition expressed to inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with an indication for SARS-CoV-2 screening
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
collection of RNA extracted nasopharyngeal and saliva samples | up to 1 month over which the samples of each participant are collected then tested
  n=130 positive n=130 negative RNA extracted from both nasopharyngeal and saliva samples from same patients sampled at the same time with suspicious COVID-19 will
collection of RNA extracted nasopharyngeal and saliva samples | up to 1 month over which the samples of each participant are collected then tested
  Collection of
  n=130 positive n=130 negative
  RNA extracted from both nasopharyngeal and saliva samples from same patients sampled at the same time with suspicious COVID-19 will enter the collection

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy M Bayette, Dr, Principal Investigator — Labosud
Locations (1):
- Bioaxiome, Nîmes, France

IPD SHARING:
Plan to Share IPD: No
the data will not be shared to other researchers since the research is an internal collection of samples; for ID SOLUTIONS